CLINICAL TRIAL: NCT05169268
Title: Real-life Assessment of Aripiprazole Long-acting Injection (Abilify Maintena) Combined With Brexpiprazole (Rexulti) in Schizophrenia: a Naturalistic Non-interventional Prospective Follow-up Study
Brief Title: Real-life Assessment of Abilify Maintena + Rexult in Schizophrenia
Acronym: MainRexult
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW-21-734
Record Dates: First submitted 2021-11-26; First posted 2021-12-23 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia and Related Disorders; Anxiety Depression
Keywords: Schizophrenia; Antipsychotics; Aripiprazole; Brexpiprazole
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; brexpiprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MainRexult Group: Subjects with schizophrenia and related disorders receiving Abilify Maintena (aripiprazole 1 monthly depot) together with Rexulti (Brexpiprazole)
  Interventions: Drug: ARIPiprazole Injection [Abilify]; Drug: Brexpiprazole

INTERVENTIONS:
Drug: ARIPiprazole Injection [Abilify] — subject already receiving the combination of Abilify Maintena and Rexulti
  Other Names: Abilify Maintena
Drug: Brexpiprazole — subject already receiving the combination of Abilify Maintena and Rexulti
  Other Names: Rexulti

SUMMARY:
MainRexult study aims to carefully evaluate a cohort of patients with schizophrenia and related disorder prescribed with the combination therapy with Abilify Maintena and Rexulti on its efficacy and tolerability in a real-life clinical setting.

DETAILED DESCRIPTION:
Currently, there is no recommendation on next-step treatment strategy if the patients remain suffering from residual symptoms, have incomplete remission, or have acute exacerbation of schizophrenia whilst receiving aripiprazole long acting injection at its recommended (maximum) dose, except to switch to other second generation antipsychotics (SGA) or to clozapine if they are in their treatment-resistant course. Such practice may incur risks of full relapse and/or unnecessary side effects to the patients, in particularly to those already showed insufficient treatment response, intolerability to side effects, or non-adherence to other antipsychotics before. On the contrary, adding another SGAs to this special cohort appears to be rational. Especially, brexpiprazole might be an ideal choice for its serotonin-dopamine activity modulator property to achieve better symptom control, and at the same time retaining the benefits from the lower incidence of side effects than other SGAs.

Cases reports on combination therapy with aripiprazole (oral or LAI) with brexpiprazole had demonstrated initial favorable outcomes, albeit lacking empirical evidence from randomized controlled trial or longer term follow-up study. Therefore, the current MainRexult study aims to carefully evaluate a cohort of patients with schizophrenia and related disorders prescribed with the combination therapy with Abilify Maintena and Rexulti on its efficacy and tolerability in an non-interventional, naturalistic real-life clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18- 65 years old at the time of enrollment
* Able to read and communicate in English and/or Chinese
* Able to give informed consent
* Has been diagnosed to have Schizophrenia (DSM-5 or ICD-10 F20 [except F20.81], Schizotypal (Personality) Disorder (DSM-5 or ICD-10 F21), or Schizoaffective Disorder (DSM-5 or ICD-10 F25), (Persistent) Delusional Disorder (DSM-5 or ICD-10 F22), Schizophreniform Disorder (DSM-5 or ICD-10 F20.81), Brief Psychotic Disorder (DSM-5) or Acute and Transient Psychotic Disorder (ICD-10 F23)
* Is receiving the combination with Abilify Maintena and brexpiprazole as treatment ≤8 weeks at the time of recruitment

Exclusion Criteria:

* Age <18 years old
* Unable to read English or Chinese
* Unable to give informed consent
* Had been diagnosed to have Intellectual Disabilities (DSM-5) or Mental Retardation (ICD-10 F70-73)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects are diagnosed with schizophrenia and related disorders who are receiving Abilify Maintena and Brexpiprazole as treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline score of the Brief Psychiatric Rating Scale-24 at 3rd and 6th months | 6 months
  Measuring efficacy on positive and negative psychotic symptoms with a total score ranges from 24 (normal) to 168 (severe ill)
Change from baseline score of the Clinical Global Impression Scale at 3rd and 6th months | 6 months
  measuring efficacy on overall clinical improvement and severity of subjects with a score ranges from 0 (normal) to 18 (severely ill)
Change from baseline score of the Hamilton Anxiety Rating Scale at 3rd and 6th months | 6 months
  measuring anxiety symptoms of the subjects with a score ranges from 0 (not ill) to 56 (severe)
Change from basline score of the Hamilton Depression Rating Scale at 3rd and 6th months | 6 months
  measuring depressive symptoms of the subjects with a score ranges from 0 (normal) to 62 (very severe)

SECONDARY OUTCOMES:
Change from basline score of the Simpson Angus Score at 3rd and 6th months | 6 months
  for intolerability assessment on extra-pyramidal side effects of the subjects from 0 (not present) to 24 (most severe)
Change from baseline score of the Barnes Akathisia Rating Scale at 3rd and 6th months | 6 months
  for intolerability assessment on akathisia of the subjects from 0 (not present) to 14 (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Albert KK Chung, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No